CLINICAL TRIAL: NCT04277819
Title: The Use of Novel Diagnostic Tools to Increase Detection of Early Fibrosis in Cystic Fibrosis Related Liver Disease to Improve Clinical Management
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00306
Record Dates: First submitted 2020-02-11; First posted 2020-02-20 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis; Liver Fibroses; Cystic Fibrosis Liver Disease
MeSH Terms: conditions — Cystic Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum is stored and will be assessed with mass spectrometry to look at blood based proteins that could be used at potential biomarkers in cystic fibrosis related liver disease
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cystic fibrosis related liver disease: Patients with cystic fibrosis, who meet the criteria for diagnosis of liver disease according to the European Cystic Fibrosis Society best practice guidelines
- Patients without cystic fibrosis related liver disease

SUMMARY:
Cystic Fibrosis (CF) is a genetic condition which affects 1 in 2500 newborn infants and is the commonest genetic condition in the UK. 1 in 25 of the white population carry the mutation. The genetic defect prevents the movement of fluids from cells, leading to thickened secretions and injury. With improvements in treatments from the commonest organ affected, the lungs, patients born with CF now can expect to live into their 40s with more than 60% living past 16.

Though better, more can be done. As treatments from lung complications have improved, the management of liver disease (second commonest organ involved) remains unchanged for a considerable time. Treatment options are limited with liver transplant the only curative option. Though potentially life-saving, it has risks and an organ shortage means alternative treatment options are desperately needed.

Identifying those with or at risk of Cystic Fibrosis related liver disease is difficult due to inadequate diagnostic tools. Routine blood tests are unreliable; therefore specific blood tests to identify scarring of the liver (biomarkers) are urgently needed. Ultrasound scan, the recommended diagnostic investigation, is only accurate in identifying the late stages of liver disease. For new therapies to be most effective we need to be able to identify patients at a much earlier stage.

This study will use multi-modality testing, including imaging techniques such as FibroScan, MRI scan and blood tests (biomarkers), to diagnose those with liver scarring and use this to better categorise disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age
2. Females will be non-pregnant and non-lactating* (for MRI scan only)
3. 20 patients with confirmed diagnosis of CF, 20 with CFLD and 20 healthy volunteers

   * Women of childbearing potential (i.e. not surgically sterilised or <1 year post menopause) will be required to:

1. Confirm they are not currently breastfeeding 2. Undergo a serum pregnancy test (serum β-HCG)

Exclusion Criteria:

1. Contraindication to magnetic resonance imaging scanning (including claustrophobia) or gadolinium-based contrast agent
2. eGFR < 50 mL/min/1.73m2
3. Pregnant or breast-feeding women.
4. Any other condition, which in the opinion of the research team may put participants at risk during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the Manchester Adult Cystic Fibrosis Centre.
  For the initial stage of the study 200 patients will be selected who are attending for their annual reviews. At this stage they will be consented, have bloods taken and FibroScan performed.
  From this initial cohort, they will be classified into presence and absence of liver disease based on current guidelines. From this 20 patients from each group along with 20 healthy volunteers will then undergo MRI scan.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Diagnostic criteria of CFLD | 2 years
  Number of participants that would be diagnosed with cystic fibrosis related liver disease according to the current European CF guidelines.
Using FibroScan as a tool to increase detection of CLFD | 2 years
  Number of participants that would be diagnosed with cystic fibrosis related liver disease with the addition of FibroScan to the diagnostic criteria
Using Biomarkers as a tool to detect CFLD | 2 years
  Number of participants with a diagnosis of CFLD that have an increase in serum biomarker values for known biomarkers of liver fibrosis.
Using MRI scan as a tool to detect CFLD | 2 years
  Number of participants with a diagnosis of CFLD that show an increase in fibrosis on their MRI scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scott JA, Jones AM, Jokl E, Gordon-Walker T, Barry PJ, Hanley NA, Piper Hanley K, Athwal VS. Improving detection of cystic fibrosis related liver disease using liver fibrosis assessment tools. Heliyon. 2023 Nov 7;9(11):e21861. doi: 10.1016/j.heliyon.2023.e21861. eCollection 2023 Nov. PMID 38053913